CLINICAL TRIAL: NCT02079207
Title: Multi-center, Randomized, Double Blinded, Phase III Trial to Assess the Immunogenicity and Safety of NBP606 in Adults 50 Years of Age and Older Who Are naïve to Pneumococcal Vaccine
Brief Title: Study Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP606_PCVA_III_2013
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBP606 (Experimental): Participants aged over 50 years are given a 0.5mL dose of 13-valent peumococcal conjugate vaccine administered on day 0.
  Interventions: Biological: NBP606
- Prodiax-23 (Active Comparator): Participants aged over 50 years are given a 0.5mL dose of 23-valent pneumococcal polysaccharide vaccine administered on day 0.
  Interventions: Biological: Prodiax-23

INTERVENTIONS:
Biological: NBP606 — 13-valent peumococcal conjugate vaccine(13vPnC)
  Arms: NBP606
Biological: Prodiax-23 — 23-valent peumococcal polysaccharide vaccine(23vPS)
  Arms: Prodiax-23

SUMMARY:
This study will assess the Immunogenicity and safety of 13-valent Pneumococcal Conjugate Vaccine compared with 23-valent Pneumococcal Polysaccharide Vaccine. All participants should be naïve of Pneumococcal vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male and Female adults over 50 years of age at screening.
* The subject who understand the requirements of the study and voluntarily consent to participate in the study.
* The subject willing to use birth control measures for the entire study duration and negative urine hCG(Human Chorionic Gonadotrophin) test at screening for women presumed to be of reproductive potential.

Exclusion Criteria:

* Known hypersensitivity to any components of the pneumococcal vaccine
* Any confirmed or suspected immunosuppressive or immunodeficient conditions including leukemia, multiple myeloma, lympoma, Hodgkin's disease, etc.
* History of autoimmune disease including multiple sclerosis(MS), lupus, polymyositis, dermatomyositis, Hashmoto's thyroiditis, Sjogren's syndrome, rheumatoid arthritis
* Functional or anatomic asplenia
* Coagulation disorder contraindicating IM(intramuscular) vaccination
* Use of any immunosuppressive therapies within the preceding 3 months including anti-cancer chemotherapies or radiation therapies and medication such as cyclophosphamide, 6-mercaptourine, azathioprine, methotrexate, steroids, cyclosporine A, rapamycin, leflunomide, TNF-α antagonist (For corticosteroids, this will mean prednisone, or equivalent dose of ≥ 15mg/day. Inhaled and topical steroids are allowed.)
* Serious chronic disorders including metastatic malignancy, severe chronic obstructive pulmonary disease requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, impaired immune function.
* Any licensed vaccine(not including diphtheria toxoid) administered within the 1 month prior to receipt of study vaccine or is scheduled to receive any other licensed vaccine(not including diphtheria toxoid) within 1 month following receipt of study vaccine.
* Subject has received diphtheria toxoid within 6 months prior to receipt of study vaccine or planned to receive diphtheria toxoid during full period of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month(Day 28) After Vaccination 1 | One month after vaccination 1
  For the comparison of OPA GMTs elicited by NBP606 relative to Prodiax-23, the 2-sided 95% CI on the geometric mean ratio(GMR) for each serotype is calculated.

SECONDARY OUTCOMES:
Serotype-specific immunoglobulin(IgG) Geometric Mean Concentration (GMC) 1 Month(Day 28) After Vaccination 1 | One Month After Vaccination 1
  For the comparison of IgG GMC elicited by NBP606 relative to Prodiax-23, the 2-sided 95% CI on the geometric mean ratio(GMR) for each serotype is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: MYUNGDON OH, MD, Study Chair — Seoul National University Hospital